CLINICAL TRIAL: NCT05973227
Title: InTRaoperative Imaging DEvice Based on endogeNous opTical Properties to Evaluate Bowel Oxygenation in Colorectal Resections: Observational First-in-human Pilot Safety Trial -TRIDENT-
Brief Title: InTRaoperative Imaging DEvice Based on endogeNous opTical Properties to Evaluate Bowel Oxygenation in Colorectal Resections
Acronym: TRIDENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1094572-01C
Record Dates: First submitted 2023-07-26; First posted 2023-08-02 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Left-sided Colorectal Resection : Diverticular Diseases; Left-sided Colorectal Resection : Colonic Neoplasms; Left-sided Colorectal Resection : Rectal Neoplasms
Keywords: Colorectal surgery; TRIDENT system; Tissue oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interventional arm (use of TRIDENT system) (Experimental)
  Interventions: Device: use of the TRIDENT system

INTERVENTIONS:
Device: use of the TRIDENT system — usage of Trident System v1.0, just before the final resection, to obtain some images of the tissue oxygenation.

SUMMARY:
The objective of the study is to assess the safety and technical feasibility of a new imaging system, used during colorectal resection surgery, named Trident in version 1.0, which could be used by the surgeon during colorectal procedures to obtain information on intestinal tissue oxygenation.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, single center, feasibility trial. All consecutive patients that fulfil the inclusion/exclusion criteria will be informed about the possibility to be included in the present clinical investigation. Only subjects that have signed the study informed consent will be included in the study. The Trident System v1.0 will be used only during approximately 2 to 5 minutes during a precise surgical step, i.e., just before the final resection of the surgical specimen. Patients will be prospectively followed at 30 days post-surgery. Data will be collected prospectively from the medical records.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for a left-sided colorectal resection, irrespective of the surgical approach (open surgery, laparoscopic surgery,) because of:

  * Colon cancer OR
  * Sigmoid diverticular disease OR
  * Rectal cancer
* All genders
* Age > 18 years old
* Ability to understand the information related to the study protocol

Exclusion Criteria:

* Pregnancy or breastfeeding
* Contraindications to anaesthesia
* Inability to provide a written informed consent
* Inclusion in a different ongoing clinical trial
* Emergency procedure
* Abdomino-perineal resection
* Hartmann procedure
* Patient is part of vulnerable population (e.g., prisoners, mentally disabled)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
image quality (sharpness, brightness, etc) and surgeon's feedback regarding the ergonomics and safety of Trident System v1.0 during surgery. | 30 days FU
  descriptive analysis on the quality images by the engineering design team and feedback provided by clinical experts (surgeons) according to ad hoc form evaluating: 1) ergonomics aspects; 2) workflow; 3) risks of breaching sterility; 4) Speed of image acquisition.

SECONDARY OUTCOMES:
- level of oxygenation (StO2) of the exteriorized colon before resection with the Trident System v1.0 - the level of oxygenation (StO2) provided by the system at the site chosen by the surgeon based on the clinical evaluation. | surgery day
  Measurement of StO2 values at the resection site determined by the surgeon based on his clinical judgment and measurement of StO2 levels over the entire length of the colon exteriorized and visible in the field of view of the Trident System v1.0.

CONTACTS AND LOCATIONS:
Overall Officials: Didier Mutter, MD, PhD, Principal Investigator — CHU Strasbourg
Locations (1):
- CHU Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No